# **Treatment Protocol: HGT-REP-081**

**Study Title:** A Multicenter Open-Label Treatment Protocol to Observe the Safety

of Replagal® (agalsidase alfa) Enzyme Replacement Therapy in

Canadian Patients with Fabry Disease

Study Number: HGT-REP-081
Study Phase: Phase III/IV

**Product Name:** Replagal (agalsidase alfa)

**Indication:** Fabry Disease **Investigators:** Multicenter

**Sponsor:** Shire Human Genetic Therapies, Inc. (Shire HGT)

**Sponsor** 700 Main Street

Contact: Cambridge, MA 02139, USA

PPD

Medical

PPD , MD

Monitor:

| | Date |
|---------------------|-------------------|
| Original Protocol: | 30 September 2010 |
| Amendment 1: | 23 November 2010 |
| <b>Amendment 2:</b> | 06 December 2010 |

# **Confidentiality Statement**

This document is the proprietary and confidential property of Shire Human Genetic Therapies, Inc.

#### **SYNOPSIS**

#### **Sponsor:**

Shire Human Genetic Therapies, Inc.

Name of Finished Product: Replagal®

Name of Active Ingredient: agalsidase alfa

**Study Title:** 

A Multicenter Open-Label Treatment Protocol to Observe the Safety of Replagal<sup>®</sup> (agalsidase alfa) Enzyme Replacement Therapy in Canadian Patients with Fabry Disease

**Study Number:** HGT-REP-081

Study Phase: Phase III/IV

Objective(s):

The objective of this study is to observe the safety of Replagal in Canadian patients with Fabry disease.

# **Study Design:**

A minimum of 60 patients and up to 150 patients are expected to participate in this treatment protocol. Patients may begin to enroll in the treatment protocol as soon as the eligibility criteria are fulfilled and informed consent is signed.

All eligible patients may receive Replagal produced by the bioreactor process (AF Replagal) on this treatment plan until AF Replagal is commercially available for the patient, the patient's participation is discontinued, or the study is discontinued, whichever comes first. Safety data will be collected throughout the treatment protocol.

#### **Population:**

The study population consists of Canadian patients with Fabry disease.

#### Test Product, Dose, and Mode of Administration:

Replagal, at a dose of 0.2 mg/kg body weight, administered by an intravenous (IV) infusion over 40 minutes, every other week (EOW)

#### **Duration of Treatment:**

Dosing will continue until AF Replagal is commercially available to the patient, the patient's participation is discontinued, or the study is discontinued, whichever comes first.

# **Efficacy Assessments:**

Not applicable

# **Safety Assessments:**

Safety endpoints, including adverse events (AEs), vital signs, blood tests, and antibodies to agalsidase alfa, will be assessed throughout this study.

#### **Statistical Methods:**

No formal statistical tests will be conducted. Tabular summaries of patient baseline demographic and clinical characteristics, patient disposition, medical history, physical examination, vital signs, adverse events, blood tests, anti-agalsidase alfa antibody, and infusion information will be produced for the safety population. The safety population includes all patients who receive at least one full or partial infusion of Replagal.

Adverse event tabular summaries will be based on all treatment-emergent adverse events recorded; AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary.

**Date of Original Approved Protocol:** 30 September 2010 **Date of Amendment 2 Approval:** 06 December 2010

# TABLE OF CONTENTS

| SY | /NOPS | IS | 2 |
|---|---|---|---|
| LI | ST OF | APPENDICES | 6 |
| LI | ST OF | ABBREVIATIONS AND DEFINITIONS OF TERMS | 7 |
| 1 | INT | RODUCTION | 9 |
| | 1.1 | Overview of Fabry Disease | 9 |
| | 1.2 | Nonclinical Studies | .10 |
| | 1.3 | Previous Human Experience | .10 |
| | 1.4 | Current Therapies | .11 |
| | 1.4 | 4.1 Replagal (agalsidase alfa) | .11 |
| | 1.4 | 4.2 Differences Between Replagal and Fabrazyme Enzyme Replacement Therapies | .12 |
| | 1.4 | 4.3 Summary of Known and Potential Risks and Benefits to Human Subjects | 12 |
| | 1.5 | Rationale | .12 |
| 2 | OBJ | ECTIVE | .13 |
| 3 | OVE | RALL DESIGN AND PLAN | .14 |
| 4 | POP | ULATION SELECTION | .15 |
| 5 | STU | DY TREATMENT(S) | .16 |
| | 5.1 | Description of Treatment(s) | .16 |
| | 5.2 | Treatment Administration | .16 |
| | 5.3 | Selection and Timing of Dose for Each Patient. | .16 |
| | 5.4 | Method of Assigning Patients to Treatment Groups. | .16 |
| | 5.5 | Blinding | .16 |
| | 5.6 | Packaging and Labeling. | .16 |
| | 5.7 | Storage | .17 |
| | 5.8 | Investigational Product Accountability and Destruction | .17 |
| 6 | TRE | ATMENT PROTOCOL PROCEDURES | .18 |
| | 6.1 | Eligibility Criteria | .18 |
| | 6.2 | Disease and Treatment History | .18 |
| | 6.3 | Demographics | .18 |
| | 6.4 | Medical History | .18 |
| | 6.5 | Physical Examination. | .19 |
| | 6.6 | Vital Signs. | .19 |
| | 6.7 | Blood Tests | .19 |
| | 6.8 | Antibody Assessments | .19 |
| | 6.9 | Replagal Administration | .20 |
| | 6.10 | Adverse Events Assessments | .20 |

# Replagal® (agalsidase alfa) Treatment Protocol HGT-REP-081 Amendment 2

| | 6. | 10.1 Definitions | |
|---|---|---|---|
| | | 6.10.1.1 Adverse Event Definition | |
| | | 6.10.1.2 Infusion-related Adverse Event Definition | |
| | | 10.2 Performing Adverse Events Assessments | |
| | | 10.3 Timing of Adverse Event Assessments | |
| | | 10.4 Relationship and Severity | |
| | | 10.5 Clarification Between Serious and Severe Adverse Events | |
| | 6. | 10.6 Protocol Deviations for Medical Emergency or Adverse Events | 22 |
| | 6.11 | Management of Infusion-related Adverse Events | 23 |
| | 6.12 | Serious Adverse Events | |
| | 6. | 12.1 Definition | 23 |
| | 6. | 12.2 Reporting Serious Adverse Events | 23 |
| | 6.13 | Pregnancy | 25 |
| | 6.14 | Removal of Patients from the Study | 25 |
| | 6.15 | Institutional Review Board /Independent Ethics Committee /Research Ethic Board (REB) | |
| | 6.16 | Ethical Conduct of the Study | |
| | 6.17 | Patient Information and Informed Consent. | |
| | 6.18 | Patient Confidentiality | |
| | 6.19 | Case Report Form Completion | |
| | 6.20 | Monitoring | |
| | 6.21 | Regulatory Administration | |
| | 6.22 | Premature Closure of the Treatment Protocol | |
| | | 22.1 Treatment Protocol Termination | |
| | | 22.2 Site Termination. | |
| | 6.23 | Record Retention | |
| | 6.24 | Publication and Disclosure Policy | |
| 7 | | TISTICAL METHODS | |
| | 7.1 | Demographic and Clinical Characteristics | |
| | 7.2 | Patient Disposition | |
| | 7.3 | Treatment Exposure | |
| | 7.4 | Anti-agalsidase alfa Antibodies | |
| | 7.5 | Adverse Events and Other Safety Assessments | |
| 8 | | ERENCES | |

# LIST OF APPENDICES

| Appendix 1 | Schedule of Events | 33 |
|------------|-----------------------------------------------------|----|
| Appendix 2 | Investigator's Signature | 34 |
| Appendix 3 | Justification for Amendments and Summary of Changes | |

#### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE adverse event

AF Replagal Replagal manufactured using the animal-component-free, bioreactor

process (agalAF1)

CFDI Canadian Fabry Disease Initiative

cGMP current Good Manufacturing Practice

CRF/eCRF case report form/electronic case report form

CRO contract research organization

ECG electrocardiogram

ELISA enzyme-linked immunosorbent assay

EOW every other week

ERT enzyme replacement therapy

EU European Union

Gb<sub>3</sub> globotriaosylceramide

GCP good clinical practice

GLA α-galactosidase A

IB Investigator's Brochure

ICH International Conference on Harmonisation

IEC independent ethics committee

IRB institutional review board

IV intravenous

MedDRA Medical Dictionary for Regulatory Activities

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse

**Events** 

NDS New Drug Submission

pHEK primary human embryonic kidney

PK pharmacokinetic

RB roller bottle Replagal
REB research ethics board

SAE serious adverse event

Shire HGT Shire Human Genetic Therapies

sNDS Supplemental New Drug Submission

SOC system organ class

transient ischemic attacks TIAs

United Kingdom UK

United States of America USA

#### 1 INTRODUCTION

# 1.1 Overview of Fabry Disease

Fabry disease is a rare, progressive, debilitating, glycosphingolipid storage disorder. It is caused by deficient activity of the lysosomal enzyme  $\alpha$ -galactosidase A which results from a mutation in the  $\alpha$ -galactosidase A gene (GLA), located on chromosome Xq22.1.  $\alpha$ -galactosidase A cleaves galactose in the alfa-anomeric configuration from glycosphingolipids, in particular globotriaosylceramide (Gb<sub>3</sub>). Mutations in the GLA gene lead to decreased or complete absence of enzyme activity that, in turn, result in accumulation of varying amounts of Gb<sub>3</sub> in cells in vascular beds, cardiomyocytes and various other cells, tissues and organs throughout the body. The clinical manifestations of Fabry disease typically include angiokeratomas, acroparesthesias, anhydrosis, anhedonia, chronic renal insufficiency leading to renal failure, hypertrophic cardiomyopathy with arrhythmias and infarction, and microvascular cerebral events including transient ischemic attacks (TIAs), stroke, and dolychoectasia. In general, patients with complete absence of  $\alpha$ -galactosidase A have a classic phenotype with rapidly progressing renal, cardiac, and cerebrovascular events whereas patients with reduced  $\alpha$ -galactosidase A have an attenuated clinical phenotype.

Clinical onset of Fabry disease typically occurs during childhood or adolescence with recurrent episodes of severe neuropathic pain in the extremities, characteristic cutaneous lesions known as angiokeratomas, and a distinctive but asymptomatic corneal dystrophy termed cornea verticillata. Vital organs, especially the heart, kidneys and brain, are progressively affected with increasing age.<sup>4</sup>

In contrast to classical X-linked disorders, females may also be affected, presumably from biased X-linked inactivation and lack of cross-cellular correction of lyonized cells by normal cells. Females may inherit an X-linked Fabry mutation from either parent and are not asymptomatic carriers. Females account for twice the number of male patients. Clinically, manifestations in females range from mild to severe phenotypes. The onset of symptoms and age of diagnosis in females occur approximately 10 years later than in males.

Before the availability of dialysis or renal transplantation, renal complications accounted for the mortality of male Fabry patients during the fourth or fifth decade of life. Median age of death in males is 50 to 55 years of age. Death in female patients with Fabry disease is, on average, a decade or more later than in males and occurs primarily as a result of cardiac or cerebrovascular complications. 9,10

Data on the true global incidence of Fabry disease are scarce and estimates vary among  $1:117,000, \sim 1:50,000$  and  $\sim 1:4,600$  live births. Estimates suggest that the ratio of patients with the later-onset: classic phenotypes are 7:1.

The diagnosis of Fabry disease may be made in males based on low levels of plasma or leukocyte  $\alpha$ -galactosidase A activity or by the presence of a gene mutation. In females, a presumptive diagnosis of Fabry disease may be based on the presence of characteristic clinical findings which must be confirmed by genotyping.

Prior to the advent of enzyme replacement therapy (ERT) in 2001, Fabry disease was an under-diagnosed condition that was primarily recognized in males with symptoms of the classical disease severity. Women were rarely diagnosed. 12-14

#### 1.2 Nonclinical Studies

The nonclinical studies have demonstrated that agalsidase alfa is well-tolerated in acute toxicology studies in mice and rats and in multiple dosing studies in rats, rabbits, and monkeys. Toxicology studies have included a single-dose IV toxicology study in rats testing doses up to 10.0 mg/kg, (a dose that is 50-fold greater than the standard human dose of 0.2 mg/kg EOW and 25-fold greater than the maximum human dose of 0.4 mg/kg once weekly tested in clinical studies [TKT027]). Chronic toxicology studies have included 13-week and a 26-week repeated IV dose studies in rats, and a 13-week repeated IV dose study in cynomolgus monkeys where doses up to 1 mg/kg/week were tested, which was 10-fold greater than the standard human dose and 2.5-fold greater than the maximum tested human dose. None of these tests showed evidence of significant toxicity associated with agalsidase alfa. In addition, an in vitro tumorigenicity study in cultured primary human embryonic kidney (pHEK) cells was performed, and this study demonstrated that agalsidase alfa did not alter the in vitro tumorigenicity or growth rates of normal primary human embryonic kidney (pHEK) cells (Data on file).

Reproductive studies in male and female rats and female rabbits revealed no untoward effects on male or female reproductive function, histopathology of reproductive organs, or embryo-fetal development. The pharmacokinetic (PK) properties and biodistribution of agalsidase alfa in mice, rats, rabbits, and monkeys have been well characterized. Following a single IV administration, serum levels of agalsidase alfa followed a biphasic distribution in several animal species including rats and monkeys. The elimination half-lives were less than 2 hours in all species, and serum levels returned to predose values 24 hours after administration. Both the maximum serum concentration immediately after dosing and the area under the concentration time curve were approximately proportional to the administered dose in rats and monkeys. There were only minor effects on PK parameters following multiple dosing in rats and monkeys.

Biodistribution studies in rats using <sup>125</sup>I-labeled agalsidase alfa have demonstrated that significant amounts of agalsidase alfa can be found in key organs pathologically affected in Fabry disease after IV administration, in particular the kidney and heart. Single and multiple-dose pharmacodynamic studies in knockout mice have demonstrated a significant reduction in Gb<sub>3</sub> in the liver, heart, and kidney.

Further details on the nonclinical studies are provided in the Investigator's Brochure (IB).

# 1.3 Previous Human Experience

Clinical studies of agalsidase alfa have been conducted in the United States, United Kingdom, Canada, Australia, Europe, Brazil, and Japan.

The clinical development program has included 3 placebo-controlled clinical studies of 6-month dosing duration in adults (TKT003, TKT005, TKT010), and open-label maintenance studies for patients continuing from these and other studies (TKT006, TKT007, TKT011, TKT013, and TKT015).

Additionally, a study in female patients (TKT014), a study in dialysis and renal transplant patients (TKT019), and a single center, open-label, compassionate use study (TKT012) have also been performed. Three studies have been conducted in children, 2 completed (TKT023 and TKT5S001), and 1 ongoing, open-label maintenance study (TKT029). An additional study (TKT028) is ongoing in patients with left ventricular hypertrophy.

There are 3 additional studies currently ongoing: Rep001a, a Phase IV study of alternative dosing regimens for Replagal in Canadian patients with Fabry disease; HGT-REP-059, a treatment protocol to provide access to Replagal for patients with Fabry disease in the United States; and HGT-REP-060, an open-label extension study for TKT028.

Over 1000 patients have been treated worldwide with Replagal (agalsidase alfa). In total, 233 adults and 37 children received Replagal in Shire HGT-sponsored studies. Long-term safety experience for patients up to 7.5 years demonstrates that Replagal therapy has been generally well tolerated in clinical studies, as well as in commercial and compassionate use.

Additional details of these clinical studies are available in the IB.

# 1.4 Current Therapies

The current approved treatment for Fabry disease is ERT. There are 2 products in this therapeutic class: agalsidase alfa, (marketed under the trade name of Replagal® in countries outside the United States, by Shire HGT) and agalsidase beta, (Fabrazyme®; Genzyme). Both are indicated for long-term treatment in patients with a confirmed diagnosis of Fabry disease ( $\alpha$ -agalactosidase A deficiency). Currently, only agalsidase beta is approved for use within the US. Replagal is currently approved in more than 40 countries worldwide.

# 1.4.1 Replagal (agalsidase alfa)

Replagal is manufactured from agalsidase alfa using an aseptic filling process in a facility in compliance with current Good Manufacturing Practice (cGMP) regulations. Replagal is formulated as a sterile product suitable for parenteral administration. The formulation of Replagal includes sodium phosphate as a buffering agent, polysorbate 20 as a stabilizing agent, and sodium chloride as an isotonic agent.

Replagal is intended for use as ERT for patients with Fabry disease. It is anticipated that replacement of the deficient enzyme may contribute to correction of the enzymatic defect, and allow for improved metabolism of the natural substrate for the enzyme. Over time, chronic replacement of the deficient enzyme could theoretically alter the natural history of Fabry disease, with concomitant improvements in renal and cardiac function, metabolism, neuropathic pain, and quality of life.

# 1.4.2 Differences Between Replagal and Fabrazyme Enzyme Replacement Therapies

Replagal is produced by a genetically engineered continuous human cell line. Fabrazyme is produced using a Chinese hamster ovary cell line. Other differences include post-translational modification of mannose residues such as glycosylation, sialylation and phosphorylation, which can potentially influence the tissue uptake and the rate of development of antibodies to the exogenously administered enzymes. Formulation excipients may also contribute to differences in individual patient sensitivities to the treatments.

The global shortage of agalsidase beta has caused a significant number of patients (approximately 700 patients globally including 500 patients in the European Union [EU] since July 2009 by Company estimates) who were previously treated with agalsidase beta to switch to treatment with agalsidase alfa. It is realized that patients switching from one ERT to another may be under the risk of carry-over effects such as emergence of adverse events observed on prior ERT or appearance of new clinical symptomology due to cross-reacting antibodies. Safety reporting has been closely monitored. There have been no unexpected safety findings and the safety profile has remained consistent over 9 years of cumulative experience.

#### 1.4.3 Summary of Known and Potential Risks and Benefits to Human Subjects

A summary of the risks and benefits for Replagal is provided in the IB.

#### 1.5 Rationale

The original Replagal New Drug Submission (NDS) was approved in Canada in 2004, indicated for long-term treatment in patients with Fabry disease. In March 2009, Shire submitted a Supplemental NDS (sNDS) for Replagal bioreactor (agalAF1 or AF) drug substance process by implementing a bioreactor process in place of the previously employed roller bottle (RB) process and eliminating animal-sourced raw materials. There are no changes to the Replagal drug product formulation, manufacturing site, manufacturing process, and container closure. Supplies of the roller bottle Replagal (RB Replagal) are quickly dwindling in Canada, and this protocol provides a mechanism to maintain uninterrupted supply of Replagal to Canadian patients.

AF Replagal is currently approved and commercialized in more than 30 countries including all EU member states, Australia, Croatia, Israel, Switzerland, Mexico, Argentina, and Paraguay. Safety data is available from approximately 1600 patients worldwide who are receiving commercially available AF Replagal. No new safety concerns have been identified.

# 2 OBJECTIVE

The objective of this protocol is to observe the safety of Replagal in Canadian patients with Fabry disease.

# 3 OVERALL DESIGN AND PLAN

A minimum of 60 patients and up to 150 patients are expected to participate in this protocol. Patients may begin to enroll in the treatment protocol as soon as the eligibility criteria are fulfilled and informed consent is signed.

All patients may continue to receive Replagal on this treatment plan until AF Replagal is commercially available for the patient, the patient's participation or the study is discontinued, whichever comes first. Safety data will be collected throughout the treatment protocol.

#### 4 POPULATION SELECTION

The population consists of Canadian patients with Fabry disease.

Each patient must meet the following criteria to receive treatment:

- 1. The patient has a documented diagnosis of Fabry disease.
- 2. The patient is sufficiently compliant with study activities to participate in this treatment plan, as judged by the Investigator.
- 3. The patient must meet current Canadian guidelines for enzyme replacement therapy for Fabry disease by having one of the following:
  - a. Age-adjusted GFR <80 mL/min or a decline in GFR of >10% which is sustained for 3 months and for which other causes of declining renal function have been excluded by a nephrologist.
  - b. Evidence of cardiac involvement related to Fabry disease including cardiac hypertrophy, valvular disease, or conduction system abnormalities.
  - c. Stroke or TIA prior to the age of 65 (documented by a neurologist) or unexplained progressive white matter changes consistent with microvascular changes on magnetic resonance imaging.
  - d. Chronic, intractable diarrhea and/or abdominal pain/cramps, refractory to standard management for at least 1 year.
  - e. Chronic, intractable neuropathic pain, refractory to analgesics and standard pain management for at least 1 year.

Patients who meet any of the following criteria will be excluded from the study:

- 1. The patient has experienced an anaphylactic or anaphylactoid reaction or other infusion-related reaction which, in the opinion of the Investigator, precludes further treatment with Replagal or may interfere with the interpretation of the study.
- 2. The patient is otherwise unsuitable for the study, in the opinion of the Investigator.

# 5 STUDY TREATMENT(S)

# **5.1** Description of Treatment(s)

All patients in this study will receive Replagal at a dose of 0.2 mg/kg body weight administered as an IV infusion over 40 minutes EOW (±5 days). Refer to the Pharmacy Manual for detailed instructions on special precautions and handling.

#### **5.2** Treatment Administration

Replagal will be provided by Shire HGT in vials as a concentrate for solution for infusion.

Replagal infusions may occur at the clinical site at home or at a qualified satellite treatment center at the investigator's discretion. Patients experiencing an infusion-related AE must receive their infusions at the clinical site until they have had 2 successive infusions without an infusion-related adverse event. Patients receiving Replagal as home therapy are required to return to the clinical site for biannual safety visits as indicated in the schedule of events (Appendix 1).

The qualified, trained medical personnel will follow the Study Procedure Manual provided separately from this protocol that outlines all operating procedures to be followed for this treatment protocol including drug transport, reconstitution, and the required patient assessments before, during, and after infusion of study drug. Clinical evaluations will remain under the medical supervision of the Investigator.

# 5.3 Selection and Timing of Dose for Each Patient

Replagal will be administered at a dose of 0.2 mg/kg body weight as an IV infusion over 40 minutes EOW (±5 days).

# 5.4 Method of Assigning Patients to Treatment Groups

Not applicable.

#### 5.5 Blinding

Not applicable.

#### 5.6 Packaging and Labeling

Replagal is supplied as a sterile, clear, colorless concentrate for dilution for IV infusion. Replagal will be provided in single use, 5 mL vials containing 3.5 mL of concentrate at a concentration of 1 mg/mL.

Study drug labels will contain information necessary to meet the applicable regulatory requirements.

# 5.7 Storage

Replagal will be provided by the Sponsor (or designee) to the clinical study sites in a temperature controlled, monitored container. The vials should be stored in a refrigerator at 2 to 8°C (36 to 46°F). A minute amount of fine particulate matter, causing the solution to appear slightly hazy, may be present during storage.

Chemical and physical in use stability can be found on the drug label.

#### 5.8 Investigational Product Accountability and Destruction

The final disposition of all investigational product delivered to an Investigator must be recorded on a patient-by-patient basis. The date and time of administration of the study drug will be documented on the appropriate case report form/electronic case report form (CRF/eCRF).

All used, partially used, and unopened study drug vials must either be returned to the Sponsor or destroyed according to Sponsor requirements.

# 6 TREATMENT PROTOCOL PROCEDURES

A complete schedule of events is provided in Appendix 1. This protocol is intended to follow the same schedule and assessments as the Canadian Fabry Disease Initiative (CFDI) protocol, and the safety visits in this protocol are intended to coincide with the twice annual visits recommended by the CFDI.

Patients enrolled in this study must be treated in accordance with current Canadian guidelines for the treatment of Fabry disease. These guidelines are provided at the following web site: www/cihr-irsc.gc.ca/e/39587.html.

# 6.1 Eligibility Criteria

Eligibility criteria (provided in Section 4) will be reviewed, and patient eligibility will be determined prior to the patient receiving the first dose of Replagal.

# **6.2** Disease and Treatment History

Documentation of diagnosis with Fabry disease will be collected up to 6 months prior to the patient receiving the first dose of Replagal.

# 6.3 Demographics

Patient demographics, including patient sex, age, and race, will be collected.

# **6.4** Medical History

A review of the patient's medical history will occur up to 6 months prior to the patient receiving the first dose of Replagal. This review will include a review of body systems, documentation of current procedures, and documentation of current concomitant medication usage. In addition, the patient will be queried on the following:

- Relevant intercurrent illness and chronic disease update
- Medication use and dose (particularly those used to treat Fabry disease)
- Site of prior ERT (ie, hospital, infusion center, doctor's office, home, other)
- Disease specific review of symptoms including:
  - o Head, neck, and thyroid
  - o Eyes, ears, nose, and throat
  - Chest and lungs
  - Heart
  - Lymph nodes
  - Abdomen
  - Anorectal
  - Genitourinary
  - Skin
  - Musculoskeletal
  - Endocrine

- Neurological
- Other

#### 6.5 Physical Examination

Complete physical examinations will occur prior to the first dose of Replagal administration and during the biannual safety visits. The physical examinations will include assessments of:

- Head, neck, and thyroid
- Eyes, ears, nose, and throat
- Chest and lungs
- Heart
- Lymph nodes
- Abdomen
- Anorectal
- Genitourinary
- Skin
- Musculoskeletal
- Endocrine
- Neurological
- Height
- Weight (within 1 week of first IV Replagal infusion)
- Other

Clinically significant findings from the physical examinations are to be reported as AEs.

# 6.6 Vital Signs

Vital signs, including blood pressure, pulse, respiratory rate, and oral temperature, will be measured immediately prior to each infusion and immediately following each infusion.

#### 6.7 Blood Tests

Blood will be collected prior to the patient receiving Replagal and at the biannual safety visits for the following assessments: serum electrolytes, creatinine, glucose, urea, potassium, sodium, chloride, bicarbonate and fasting lipids profile.

# 6.8 Antibody Assessments

Blood samples will be collected for determination of anti-agalsidase alfa antibodies prior to the patient receiving Replagal and at the biannual safety visits.

Blood samples collected for anti-agalsidase antibody determination will be evaluated at Shire HGT

These samples will be screened using an enzyme-linked immunosorbent assay (ELISA).

Positive samples will be isotyped (IgG, IgA, IgM, or IgE). In addition, positive samples will be tested for enzyme neutralizing activity using an in vitro assay.

# 6.9 Replagal Administration

Patients will receive Replagal IV infusions EOW until Replagal is commercially available to the patient, or the patient's participation or the study is discontinued.

Replagal administration will occur as described in Section 5.2; home infusions may occur.

#### **6.10** Adverse Events Assessments

#### **6.10.1 Definitions**

#### **6.10.1.1** Adverse Event Definition

An adverse event (AE) is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, and/or laboratory changes occurring in any phase of a clinical study, and whether or not considered study drug-related. This includes an exacerbation of a pre-existing condition. Adverse events will be collected from informed consent until 30 days after the last dose of study drug and/or until the event has been resolved/stabilized or an outcome is reached, whichever comes first. For patients who discontinue or are withdrawn, AEs will be followed up to 30 days after their last infusion of Replagal.

Adverse events include:

- Worsening (change in nature, severity, or frequency) of conditions present at the onset of the treatment plan
- Intercurrent illnesses
- Drug interactions
- Abnormal laboratory values (this includes significant shifts within the range of normal that the Investigator considers to be clinically important)
- Clinically significant abnormalities in physical examination, vital signs, and weight

Throughout the treatment protocol, the Investigator must record all AEs on the AE CRF/eCRF, regardless of the severity or relationship to study drug. The Investigator should treat patients with AEs appropriately and observe them at suitable intervals until the events stabilize or resolve. Adverse events may be discovered through observation or examination of the patient, questioning of the patient, complaint by the patient, or by abnormal clinical laboratory values, or abnormal electrocardiogram (ECG).

In addition, AEs may also include unexpected laboratory values that become significantly out-of-range and determined to be clinically significant by the Investigator.

In the event of an unexpected out-of-range value, the laboratory test should be repeated until it returns to normal or can be explained and the patient's safety is not at risk.

#### 6.10.1.2 Infusion-related Adverse Event Definition

An infusion-related adverse event will be defined as an adverse event that 1) begins either during or within 12 hours after the start of the infusion, and 2) is judged as possibly or probably related to study drug. Infusion-related adverse events are to be managed as defined in Section 6.11.

#### **6.10.2** Performing Adverse Events Assessments

Patients should be asked non-leading questions, eg, "How do you feel?" and further questions should be posed if there is indication of an AE. The questioning should be conducted with due regard for objectivity and, in particular, the questioner should gather information regarding AEs from questioning the patient, spontaneous reporting by the patient, laboratory reports, and any health care provider's observations.

The onset date, resolution date, treatment administered, and outcome of each AE must be recorded on the appropriate CRF. In addition, the relationship of each AE to study drug must be recorded.

#### **6.10.3** Timing of Adverse Event Assessments

Adverse events will be assessed from the time the patient provides signed informed consent until 30 days after the patient's final infusion of Replagal on this treatment plan. The final AE assessment may be performed at the clinical site or by telephone call.

# 6.10.4 Relationship and Severity

The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0 grading scale should be referenced when assessing the severity of an AE. If an AE is not described in the NCI CTCAE v3.0, the severity should be recorded based on the scale below. The severity of all AEs/SAEs should be recorded on the appropriate CRF/eCRF page as Grade 1, 2, 3, or 4 corresponding, respectively, to a severity of mild, moderate, severe, or life-threatening.

# Relationship to Product(s) Definition

| 1 () | |
|---|---|
| Not Related | Unrelated to study drug. |
| Possibly Related | A clinical event/laboratory abnormality with a reasonable time sequence to administration of study drug, but which could also be explained by concurrent disease or other drugs/chemicals. |
| Probably Related | A clinical event/laboratory abnormality with a reasonable time sequence to administration of study drug, unlikely to |

| Relationship to Product(s) | Definition |
|---|---|
| | be attributable to concurrent disease or other drugs and chemicals and which follows a clinically reasonable response on de-challenge. |
| | The association of the clinical event/laboratory abnormality must also have some biologic plausibility, at least on theoretical grounds. |

| AE Severity | Definition |
|----------------------------|------------------------------------------|
| Grade 1 (Mild) | No limitation of usual activities. |
| Grade 2 (Moderate) | Some limitation of usual activities. |
| Grade 3 (Severe) | Inability to carry out usual activities. |
| Grade 4 (Life-threatening) | Immediate risk of death. |

#### 6.10.5 Clarification Between Serious and Severe Adverse Events

The term "severe" is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This is not the same as "serious," which is based on the outcome or action criteria usually associated with events that pose a threat to life or functioning. Seriousness (not severity) and causality serve as a guide for defining regulatory reporting obligations.

# 6.10.6 Protocol Deviations for Medical Emergency or Adverse Events

During and following a patient's participation in the treatment protocol, the Investigator should ensure that adequate medical care is provided to a patient for any AEs, including clinically significant laboratory test results. The Investigator should inform the patient, the patient's parent(s), or the patient's legally authorized representative when medical care is needed for intercurrent illness(es) of which the Investigator becomes aware. In an emergency situation, the Investigator should contact the Shire HGT Medical Monitor.

Only when an emergency occurs that requires an immediate deviation from the protocol for the safety of a patient, will there be such a deviation, and this will be only for that patient. The Investigator or other physician in attendance in such an emergency must contact the Shire HGT Medical Monitor as soon as possible. The Investigator, along with the Shire HGT Medical Monitor, will make a decision as to whether or not the patient should continue in the treatment protocol. The departure from the protocol and the grounds for it should be stated in the CRF.

# 6.11 Management of Infusion-related Adverse Events

If a patient has an infusion-related adverse event during the infusion of study drug, the Investigator should decide, based on his or her clinical judgment, whether the infusion should be slowed, or temporarily or permanently discontinued. Infusion-related adverse events that occur post-infusion should be assessed and treated in a similar manner.

Patients experiencing a recurrent infusion-related adverse event may be premedicated. If infusions continue without incident, then tapering of medications can be considered.

In case of severe infusion-related adverse events, the Investigator should consult with the Shire HGT Medical Monitor prior to the patient's next dose to determine the appropriate course of action for future infusions.

#### **6.12 Serious Adverse Events**

#### 6.12.1 Definition

A serious adverse event (SAE) is defined by federal regulation as any AE occurring at any dose that results in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect.

Important medical events that may not result in death, be life threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

Hospitalizations, which are the result of elective or previously scheduled surgery for preexisting conditions, which have not worsened after initiation of treatment, should not be classified as SAEs. For example, an admission for a previously scheduled ventral hernia repair would not be classified as an SAE. If however complications were to develop they would be evaluated to determine if serious criteria had been met.

# **6.12.2** Reporting Serious Adverse Events

Any SAE, regardless of relationship to study medication and which occurs in a patient after informed consent is obtained, should be recorded by the clinical site on a SAE form that is to be transmitted to the Shire HGT Medical Monitor and Shire's Global Pharmacovigilance Department at the fax contact number provided below. The SAE must be completely described on the patient's CRF/eCRF, including the judgment of the Investigator as to the relationship of the SAE to the study drug. The Investigator will promptly supply all information identified and requested by Shire HGT (and/or contract research organization [CRO]) regarding the SAE. The Investigator must report the SAE to Shire Global Pharmacovigilance and to the Shire HGT Medical Monitor on a SAE form.

This form must be completed and FAXED within 24 hours of the Investigator learning of the event to:

Fax SAE Form to

Shire Pharmacovigilance and Risk Management Department:

International FAX: PPD (UK) OR United States FAX:

PPD

And

Telephone: PPD or PPD

AND

Shire HGT Medical Monitor: FAX PPD (USA)

Any follow-up information must also be completed on a SAE form and faxed to the same numbers listed above.

In the event of a severe, unexpected, fatal or life-threatening and possibly or probably related SAE, the clinical site should complete the SAE form and transmit the SAE form to the Shire HGT Medical Monitor and to Shire's Global Pharmacovigilance Department (as stated above) within 24 hours. In addition, the clinical site must contact the Shire HGT Medical Monitor or the Shire Global Pharmacovigilance Department immediately by telephone or e-mail. The following provides contact information for the Shire Global Pharmacovigilance Department and the Shire HGT Medical Monitor.

If an SAE is assessed as severe or life-threatening and possibly/probably related, contact by phone:



In the event that the Shire's Global Pharmacovigilance Department and the Shire HGT Medical Monitor cannot be reached, a message and fax must be left at the emergency numbers listed above within 24 hours of the incident.

The Investigator must promptly report in a timely manner to his/her IRB/IEC/REB, all SAEs and any unanticipated problems involving risk to human patients. It is the responsibility of Shire HGT to ensure that each Investigator receives a copy of any CIOMS I/Med Watch report that has been submitted to the appropriate regulatory agency(ies) notifying them of a related SAE/SUSAR. The Investigator or Shire HGT must ensure that the IRB/IEC/REB receives a copy of the report and that a copy is also filed within their study files. In addition, Shire HGT will also notify the Investigators and IRBs/IECs/REBs of any deaths occurring during the treatment protocol.

# 6.13 Pregnancy

The Sponsor must be notified in the event of a pregnancy occurring during the course of the study and through 30 days after the patient's last dose of study drug. Pregnancy is not to be reported as an AE; the pregnancy form should be used to report the pregnancy. The pregnancy will be followed through delivery or final outcome.

# 6.14 Removal of Patients from the Study

Patients may withdraw from the treatment protocol at any time. The Investigator or Sponsor may withdraw a patient from the treatment protocol for the following medical or administrative reasons:

- Adverse Event: If a patient experiences an AE which, in the judgment of the Investigator, the Sponsor, or the Shire HGT Medical Monitor, presents an unacceptable consequence or risk to the patient, the patient will be withdrawn from the treatment protocol.
- Adverse Laboratory Experience: If a patient has an adverse laboratory experience which, in the judgment of the Investigator, the Sponsor, or the Shire HGT Medical Monitor, presents an unacceptable consequence or risk to the patient, the patient will be withdrawn from the treatment protocol.
- Comorbidity: If a patient develops a comorbidity during the course of the treatment protocol that is not associated with the condition under study, and which requires treatment that is not consistent with protocol requirements, the patient will be withdrawn from the treatment protocol. A patient will be withdrawn from the treatment protocol if, in the judgment of the Investigator, s/he develops an intercurrent illness that, in any way, justifies his withdrawal.
- Refusal of Treatment: If for any reason the patient refuses treatment during the treatment protocol, the patient will be withdrawn from the treatment protocol, and the reason for refusal will be documented on the CRF. Reasonable efforts will be made to monitor the patient for AEs following such discontinuation. Such efforts will be documented in the CRF.
- Withdrawal of Informed Consent: A patient may withdraw his informed consent to participate in the treatment protocol at any time and for any reason.
- Lack of Efficacy: The patient will be withdrawn from the treatment protocol if, in the opinion of the CFDI Investigator, a lack of efficacy is observed.

At the time of discontinuation or withdrawal, patients will undergo all safety and efficacy evaluations required for the End of Study visit. The Investigator will complete the appropriate CRF describing the reason for discontinuation.

In addition, patients who withdraw or are discontinued will have a follow-up assessment for safety at the clinical site 30 days after their last infusion of Replagal.

# 6.15 Institutional Review Board /Independent Ethics Committee /Research Ethics Board (REB)

Before initiation of the treatment protocol, the Investigator must provide the Sponsor with a copy of the written IRB/IEC/REB approval of the protocol and the informed consent form. This approval must refer to the informed consent form and to the study title, study number, and version and date of issue of treatment protocol, as given by the Sponsor on the cover page of the protocol. Local IRBs may be given the option to delegate to the central IRB identified for the study.

Status reports must be submitted to the IRB/IEC/REB at least once per year. The IRB/IEC/REB must be notified of completion of the treatment protocol. Within 3 months of treatment protocol completion or termination, a final report must be provided to the IRB/IEC/REB. A copy of these reports shall be sent to the study clinical monitor. The Investigators must maintain an accurate and complete record of all submissions made to the IRB/IEC/REB, including a list of all reports and documents submitted. Adverse events which are reported to Health Canada or other regulatory agencies must be submitted promptly to the IRB/IEC/REB.

# **6.16** Ethical Conduct of the Study

The procedures set out in this study protocol, pertaining to the conduct, evaluation, and documentation of this study, are designed to ensure that the Sponsor and Investigators abide by good clinical practice (GCP) as described in the 21 CFR Parts 50, 56, and 312 and the International Conference on Harmonisation (ICH) GCP Guidelines Compliance with these regulations and guidelines also constitutes compliance with the ethical principles described in the Declaration of Helsinki.

# 6.17 Patient Information and Informed Consent

Before enrolling in the treatment protocol, each patient, the patient's parent(s), or the patient's legally authorized representative(s) must consent to participate after the nature, scope, and possible consequences of the treatment protocol have been explained in a form understandable to him/her. An informed consent form that includes information about the treatment protocol will be prepared and given to the patient, the patient's parent(s), or the patient's legally authorized representative. This document will contain all Health Canada and ICH-required elements. The informed consent form must be in a language understandable to the patient, the patient's parent(s), or the patient's legally authorized representative(s) and must specify who informed the patient, the patient's parent(s), or the patient's legally authorized representative(s).

After reading the informed consent document, the patient, the patient's parent(s), or the patient's legally authorized representative must give consent in writing. The patient's consent must be confirmed at the time of consent by the personally dated signature of the patient, the patient's parent(s) or the patient's legally authorized representative and by the personally dated signature of the person conducting the informed consent discussions.

If the patient, the patient's parent(s), or the patient's legally authorized representative is unable to read, oral presentation and explanation of the written informed consent form and information to be supplied to the patient must take place in the presence of an impartial witness. Consent must be confirmed at the time of consent orally and by the personally dated signature of the patient, or by a local legally recognized alternative (eg, the patient's thumbprint or mark) or by the personally dated signature of the patient's parent(s) or the patient's legally authorized representative. The witness and the person conducting the informed consent discussions must also sign and personally date the informed consent document. It should be recorded and dated in the source document that consent was given.

A copy of the signed and dated consent document(s) must be given to the patient, the patient's parent(s), or the patient's legally authorized representative. The original signed consent document will be retained by the Investigator.

The Investigator will not undertake any measures specifically required solely for the treatment protocol until valid consent has been obtained.

A model of the informed consent form to be used in this treatment protocol will be provided to the sites separately from this protocol.

Where applicable, signed assent(s) to participate in the treatment protocol will be obtained.

### **6.18 Patient Confidentiality**

Patient names will not be supplied to the sponsor. Only the patient number and patient initials will be recorded in the CRF/eCRF, and if the patient name appears on any other document, it must be obliterated before a copy of the document is supplied to the Sponsor. Study findings stored on a computer will be stored in accordance with local data protection laws. The patients will be told that representatives of the sponsor, a designated contract research organization (CRO), the IRB/IEC/REB, or regulatory authorities may inspect their medical records to verify the information collected, and that all personal information made available for inspection will be handled in strictest confidence and in accordance with local data protection laws. The Investigator will maintain a personal patient identification list (patient numbers with the corresponding patient names) to enable records to be identified.

# **6.19 Case Report Form Completion**

Case Report Forms (paper or electronic) are provided for each patient. All forms must be filled out by authorized study personnel. All corrections to the original CRF entry must indicate the reason for change.

The Investigator is required to sign the CRF after all data have been captured for each patient. If corrections are made after review and signature by the Investigator, he or she must be made aware of the changes, and his or her awareness documented by resigning the CRF.

#### 6.20 Monitoring

Monitoring procedures that comply with current GCP guidelines will be followed. Review of the CRF's for completeness and clarity, cross-checking with source documents, and clarification of administrative matters will be performed.

The study will be monitored by the Sponsor or its designee. Monitoring will be performed by a representative of the Sponsor (Clinical Study Monitor) who will review the CRFs and source documents. The site monitor will ensure that the investigation is conducted according to protocol design and regulatory requirements by frequent site visits and communications (letter, telephone, and facsimile).

# **6.21 Regulatory Administration**

Appropriate regulatory documentation will be collected as mandated by Health Canada.

#### **6.22** Premature Closure of the Treatment Protocol

#### **6.22.1 Treatment Protocol Termination**

If the sponsor or an Investigator discovers conditions arising during the treatment protocol which indicate that the clinical investigation should be halted due to an unacceptable patient risk, the treatment protocol may be terminated after appropriate consultation between Shire HGT and the Investigators.

In addition, a decision on the part of Shire HGT to suspend or discontinue development of the test material may be made at any time.

#### **6.22.2 Site Termination**

A specific site may be terminated separate from the general treatment protocol for, but not limited to, the following conditions:

- The discovery of an unexpected, significant, or unacceptable risk to the patients enrolled at the site.
- Insufficient adherence by the Investigator to protocol or regulatory requirements.

# **6.23 Record Retention**

Essential documents should be retained by the site for at least 2 years after the last approval of a marketing application and until there is no pending or contemplated marketing applications or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. The sponsor will notify the Investigator if these documents must be retained for a longer period of time. It is the responsibility of the Sponsor to inform the Investigator/institution as to when these documents no longer need to be retained.

Records will be maintained by the Sponsor for a period of 25 years and will be accessible for onsite inspection by Health Canada inspectors.

# **6.24** Publication and Disclosure Policy

All information concerning the study material, such as patent applications, manufacturing processes, basic scientific data, and formulation information supplied by the Sponsor and not previously published are considered confidential and will remain the sole property of the Sponsor. The Investigator agrees to use this information only in accomplishing this study and will not use it for other purposes.

It is understood by the Investigator that the information developed in the clinical study may be disclosed as required to the authorized regulatory authorities and governmental agencies.

In order to allow for the use of the information derived from the clinical studies, it is understood that there is an obligation to provide the Sponsor with complete test results and all data developed in the study in a timely manner.

The Investigator and any other clinical personnel associated with this study will not publish the results of the study, in whole or in part, at any time, unless they have consulted with Shire HGT, provided Shire HGT a copy of the draft document intended for publication, and obtained Shire HGT's written consent for such publication. All information obtained during the conduct of this study will be regarded as confidential. Shire HGT will use the information for registration purposes and for the general development of the drug.

#### 7 STATISTICAL METHODS

No formal statistical tests will be conducted. Tabular summaries of patient baseline demographic and clinical characteristics, patient disposition, medical history, physical examination, vital signs, adverse events, anti-agalsidase alfa antibody, and infusion information will be produced for the safety population. The safety population includes all patients who receive at least one full or partial infusion of Replagal. Continuous data collected prior to receiving study drug and at subsequent visits will be summarized using descriptive statistics (n, mean, median, minimum, maximum, and standard deviation). Categorical data will be summarized as frequencies and percentages.

# 7.1 Demographic and Clinical Characteristics

Baseline demographics and other patient characteristics, including disease history, physical exam, vital signs, and medical history will be presented.

# 7.2 Patient Disposition

The disposition of all enrolled patients will be summarized with frequencies and percentages including patients who completed the study and patient who discontinued study treatment prior to the end of study visit.

# 7.3 Treatment Exposure

Infusion information will be listed by patient and visit. The cumulative dose of study drug taken, and the duration of study drug exposure will be summarized descriptively.

# 7.4 Anti-agalsidase alfa Antibodies

Antibody data will be listed by patient and visit. The status of antibodies and neutralizing antibody will be summarized descriptively.

#### 7.5 Adverse Events and Other Safety Assessments

Adverse event tabular summaries will be based on all treatment-emergent adverse events recorded; AEs will be coded using the MedDRA coding dictionary.

AEs will be summarized by system organ class (SOC) and preferred term. The total number of AEs by SOC and preferred term, as well as the number and proportion of patients experiencing an AE will be tabulated; a patient will be counted only once within each SOC and preferred term. AEs by SOC and preferred term will be tabulated by severity. In the case of multiple occurrences of the same AEs (at the preferred term level) in an individual patient, the AE that is classified as the most severe (ie, maximum severity) will be identified for the analysis by severity. In addition, AEs by SOC and preferred term will be tabulated by relationship to study drug by reporting the episode with the closest relationship to study drug.

The number and percentage of patients reporting serious adverse events will be presented by SOC and preferred term; in addition, an SAE listing will be presented.

The number and percentage of patients reporting an infusion-related adverse event will be presented by SOC and preferred term. An infusion-related adverse event is defined as an AE that: (1) begins either during or within 12 hours after the start of the infusion, and (2) is judged by the investigator to be possibly or probably related to study drug.

The number and proportion of patients experiencing an AE(s) that led to permanent discontinuation will be summarized by SOC and preferred term. Furthermore, a listing of all patients who permanently discontinued due to an AE(s) will be provided.

Furthermore, safety will be evaluated by assessing vital signs and blood tests. Data for vital signs and blood tests will be listed for each patient and abnormal values will be flagged. Shift tables from baseline to last visit may be presented for vital signs, and a summary table may be presented for blood tests.

#### 8 REFERENCES

- 1. Garman SC, Garboczi DN. The molecular defect leading to Fabry disease: structure of human alpha-galactosidase. J Mol Biol 2004;337(2):319-35.
- 2. Schiffmann R, Ries M. Fabry's disease--an important risk factor for stroke. Lancet 2005;366(9499):1754-6.
- 3. Ries M, Kim HJ, Zalewski CK, et al. Neuropathic and cerebrovascular correlates of hearing loss in Fabry disease. Brain 2007;130(Pt 1):143-50.
- 4. Ries M, Gupta S, Moore DF, et al. Pediatric Fabry disease. Pediatrics 2005;115(3):e344-55.
- 5. Ries M, Ramaswami U, Parini R, et al. The early clinical phenotype of Fabry disease: a study on 35 European children and adolescents. Eur J Pediatr 2003;162(11):767-72.
- 6. Eng CM, Fletcher J, Wilcox WR, et al. Fabry disease: baseline medical characteristics of a cohort of 1765 males and females in the Fabry Registry. J Inherit Metab Dis 2007;30(2):184-92.
- 7. Deegan PB, Baehner AF, Barba Romero MA, Hughes DA, Kampmann C, Beck M. Natural history of Fabry disease in females in the Fabry Outcome Survey. J Med Genet 2006;43(4):347-52.
- 8. MacDermot KD, Holmes A, Miners AH. Anderson-Fabry disease: clinical manifestations and impact of disease in a cohort of 98 hemizygous males. J Med Genet 2001;38(11):750-60.
- 9. MacDermot KD, Holmes A, Miners AH. Anderson-Fabry disease: clinical manifestations and impact of disease in a cohort of 60 obligate carrier females. J Med Genet 2001;38(11):769-75.
- 10. Gupta S, Ries M, Kotsopoulos S, Schiffmann R. The relationship of vascular glycolipid storage to clinical manifestations of Fabry disease: a cross-sectional study of a large cohort of clinically affected heterozygous women. Medicine (Baltimore) 2005;84(5):261-8.
- 11. Meikle PJ, Hopwood JJ, Clague AE, Carey WF. Prevalence of lysosomal storage disorders. JAMA 1999;281(3):249-54.
- 12. Spada M, Pagliardini S, Yasuda M, et al. High incidence of later-onset Fabry disease revealed by newborn screening. Am J Hum Genet 2006;79(1):31-40.
- 13. Cho ME, Kopp JB. Fabry disease in the era of enzyme replacement therapy: a renal perspective. Pediatr Nephrol 2004;19(6):583-93.
- 14. Wilcox W, Oliveira J, Hopkin R, et al. Fabry Registry. Females with Fabry disease frequently have major organ involvement: lessons from the Fabry Registry. Mol Genet Metab 2008;93(2):112-28.

# **Appendix 1 Schedule of Events**

| | Within 6 | Treatment Period | | |
|---|---|---|---|---|
| Evaluation | Months<br>Prior to<br>First Dose | Dosing Every<br>Other Week<br>(±5 days) | Biannual Visits<br>to Site <sup>a</sup> | End of Study<br>(30 days after<br>last dose) |
| Informed Consent | X | | | |
| Treatment Protocol Entry Criteria | X | | | |
| Medical History | X | | | |
| Demographics | X | | | |
| Disease and Treatment History | X | | | |
| Physical Examination <sup>b</sup> | X | | X | |
| Weight | | X <sup>e</sup> | X | |
| Vital Signs <sup>c</sup> | | X | X | |
| Blood Tests <sup>d</sup> | X | | X | |
| Serum Anti-agalsidase alfa<br>Antibody | X | | X | |
| Drug Administration | | X | X | |
| AE Assessment | | X | X | X |

Abbreviations: AE = adverse event; CFDI = Canadian Fabry Disease Initiative

- Biannual visits are intended to coincide with visits in the Canadian Fabry Disease Initiative (CFDI) protocol. Procedures and study assessments during these visits will be performed at the clinical site. For patients receiving home infusions, the infusions given at the biannual visits may be administered at the clinical site.
- Physical examination includes assessments of head, neck, and thyroid; eyes, ears, nose, and throat; chest and lungs; heart; lymph nodes; abdomen; anorectal; genitourinary; skin; musculoskeletal; endocrine; neurological; height; weight; and other.
- Include blood pressure, pulse, respiratory rate, and oral temperature. Vitals signs are taken immediately before and immediately after every infusion.
- Includes serum electrolytes, creatinine, glucose, urea, potassium, sodium, chloride, bicarbonate and fasting lipids profile.
- Subject weight should be obtained prior to the Week 1 infusion

| Appendix 2 | Investigator's Signature | |
|---|---|---|
| Study Title: | A Multicenter Open-Label Treatment Protocol to Observe the Safety of Replagal® (agalsidase alfa) Enzyme Replacement Therapy in Canadian Patients with Fabry Disease | |
| <b>Study Number:</b> | HGT-REP-081 | |
| Final Date<br>Amendment 2: | 6 December 2010 | |
| I have read Study I conduct the study a | | nvestigator's Brochure, and I agree to |
| Signatory | | |
| Investigator | Signature | Date |
| | Print Name | Institution |
| Shire HGT<br>Medical | | |
| Monitor | Signature | Date |
| | Print Name | |

# **Appendix 3 Justification for Amendments and Summary of Changes**

# **Amendment 1:**

The protocol was submitted to Health Canada on 8 October 2010 as part of a Treatment Use Clinical Trial Application. The Agency requested several changes and additions to the protocol (Clarifax 2 November 2010) and the changes proposed by Shire were approved by the Agency, on 4 November 2010. The amendment incorporates changes that address comments received from the Agency.

Changes to the amendment are detailed below. New text is indicated as bold font, and deleted text is indicated as strikethrough.

#### Section 3: Overall Design and Plan

Health Canada requested that a minimum number of patients be specified in order to obtain meaningful safety data from this safety clinical trial. Shire plans to include a minimum number of 60 patients. With a minimum of 60 subjects, there will be at least a 95% chance of observing at least one AE of a given type, if the event has a frequency of 5%.

The amended text reads as follows:

Approximately 150 patients are expected to participate in this treatment protocol, although the number may be increased or decreased depending upon patient need or patient availability A minimum of 60 patients and up to 150 patients are expected to participate in this protocol. Patients may begin to enroll in the treatment protocol as soon as the eligibility criteria are fulfilled and informed consent is signed.

Other sections affected by this change: Synopsis

#### **Section 4: Population Selection**

Health Canada requested that the following be added as exclusion criteria.

#### Patients who meet any of the following criteria will be excluded from the study:

- 1. The patient has experienced an anaphylactic or anaphylactoid reaction or other infusion-related reaction which, in the opinion of the Investigator, precludes further treatment with Replagal or may interfere with the interpretation of the study
- 2. The patient is otherwise unsuitable for the study, in the opinion of the Investigator.

Other sections affected by this change: None

#### **Section 6.2: Disease and Treatment History**

The screening period for the study has been clarified. Screening data will be obtained during the 6 months prior to the patient's initiation of treatment with Replagal, to align with the patients' current biannual assessment schedule in the CFDI. The added text reads:

Documentation of diagnosis with Fabry disease will be collected **up to 6 months** prior to the patient receiving the first dose of Replagal.

Other sections affected by this change: Section 6.4, Medical History; Appendix 1, Schedule of Events

#### **Section 6.14: Removal of Patients from Study Drug**

Health Canada requested that "lack of efficacy" be included as a criterion for withdrawal from the study.

The added text is the last bullet in the list:

• Lack of Efficacy: The patient will be withdrawn from the treatment protocol if, in the opinion of the CFDI Investigator, a lack of efficacy is observed.

Other sections affected by this change: None

#### **Amendment 2:**

The protocol was amended to address several minor inconsistencies. Also, the procedures for study monitoring were clarified.

#### 6.10.1.2 Infusion-Related Adverse Event Definition

An infusion-related adverse event will be defined as an adverse event that 1) begins either during or within 12 hours after the start of the infusion, and 2) is judged as possibly or probably related to study drug. Infusion-related adverse events are to be managed as defined in Section 6.11

#### **Section 6.20: Study Monitoring**

The text has been amended to clarify the procedures used for study monitoring.

Formerly read:

Site qualification and initiation will be completed via teleconference. Investigator site monitoring will be done remotely at up to 10% of the total number of sites with the exception of 'for cause' on site monitoring visits.

Now reads:

Monitoring procedures that comply with current Good Clinical Practice (GCP) guidelines will be followed. Review of the CRF's for completeness and clarity, cross-checking with source documents, and clarification of administrative matters will be performed.

The study will be monitored by the Sponsor or its designee. Monitoring will be performed by a representative of the Sponsor (Clinical Study Monitor) who will review the CRFs and source documents.

The site monitor will ensure that the investigation is conducted according to protocol design and regulatory requirements by frequent site visits and communications (letter, telephone, and facsimile).

Other sections affected by this change: None

# **Appendix 1:**

Subject weight is required to ensure correct dosing. The physical examination is listed with weight required at certain visits, but a separate row has been added for weight and noted that weight should also be measured during the Week 1 visit prior to the first dose of Replagal.

Other sections affected by this change: None